CLINICAL TRIAL: NCT02113930
Title: Analysis of Clinical and Immunological Characteristics, as Well as Pathophysiological Mechanisms in a French Cohort of Patients With Idiopathic CD4 Lymphocytopenia
Brief Title: Idiopathic CD4 Lymphocytopenia
Acronym: Lympho-4
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI08039
Record Dates: First submitted 2013-03-28; First posted 2014-04-15 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic CD4 Lymphocytopenia
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive | interventions — Genetic Association Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum; plasma, peripheral blood mononuclear cells and DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Idiopathic CD4 lymphocytopenia: Constitution of a biobank of frozen cells, plasma and serum samples
  Interventions: Biological: Constitution of a biobank of frozen cells, plasma and serum samples
- Genetic Study: High rate genome wide genetic screening, investigation of mutations associated with identified primary immune deficiencies (adenosine deaminase et class II MHC)
  Interventions: Genetic: Genetic study

INTERVENTIONS:
Biological: Constitution of a biobank of frozen cells, plasma and serum samples — Depending on clinical presentation and based on previous data obtained by our group, we will investigate the immune responses against Human papilloma virus (HPV), Cryptococcus neoformans,implication of chemokines involved in lymphocyte migration (CXCR4 and CCR7 receptors) and signalisation in response to cytokines controlling LT CD4+ homeostasis (IL-7 et IL-2).
  Groups: Idiopathic CD4 lymphocytopenia
Genetic: Genetic study — High rate genome wide genetic screening, investigation of mutations associated with identified primary immune deficiencies (adenosine deaminase et class II MHC)
  Groups: Genetic Study

SUMMARY:
Definition: Idiopathic CD4+ T lymphocytopenia (ICL) is an immune deficiency first described in 1992 and characterized by the US Centers for Disease Control (CDC) as absolute CD4+ T-lymphocyte count < 300/mm3 or < 20% of total T cells on more than one cell count; no evidence of infection with HIV-1/2 or human T-cell lymphotropic 1/2 (HTLV-1/2); and lack of a defined immune-deficiency disease or therapy for lymphocytopenia. Epidemiologic, clinical and immunological characteristics of the syndrome were described in 1993 and ICL is now considered a heterogeneous syndrome not caused by an infectious agent. Patients with ICL may show opportunistic infections such as disseminated Cryptococcus neoformans infection, Pneumocystis jiroveci pneumonia and John Cunningham (JC) virus infection as a result of profound cell-mediated immune-response deficiency.

Few studies have focused on the pathophysiology of ICL. CD4+ T-lymphocyte phenotyping revealed increased CD95 expression that could be responsible for excess apoptosis leading to lymphocytopenia. Moreover, the membrane expression of C-X-C chemokine receptor type 4 (CXCR4) was found impaired in T lymphocytes with ICL, and CXCR4 trafficking was improved with interleukin 2 (IL-2) treatment in some patients. Recently, mutations in nunc119, MAGT1 and Rag were found associated with CD4+ T lymphocytopenia. In a prospective study of 39 patients, CD8+ T lymphocytopenia (<180/mm3) and degree of CD4+ T-cell activation measured by human leukocyte antigen DR (HLA-DR) expression was found associated with poor prognosis.

ICL is a heterogeneous disorder often associated with deficiencies in CD8+, CD19+, and/or NK cells. Long-term prognosis may be related to initial CD4+ and NK cell deficiency.

Larger studies are needed to better identify the patients who might benefit from IL-2 therapy. This is why the investigators conduct the Lympho-4 study, in which the investigators plan to include 200 patients with a suspected/proven diagnosis of ICL.

DETAILED DESCRIPTION:
Definition. Idiopathic CD4+ T lymphocytopenia (ICL) is an immune deficiency first described in 1992 and characterized by the US Centers for Disease Control (CDC) as absolute CD4+ T-lymphocyte count < 300/mm3 or < 20% of total T cells on more than one cell count; no evidence of infection with HIV-1/2 or human T-cell lymphotropic 1/2 (HTLV-1/2); and lack of a defined immune-deficiency disease or therapy for lymphocytopenia.

ICL is a heterogeneous disorder often associated with deficiencies in CD8+, CD19+, and/or NK cells. Thus, ICL does not correspond to a unique disease but more probably to a number of different conditions with distinct underlying mechanisms. This is why the investigators decided to launch the Lympho-4 study, in which the investigators plan to include 200 patients with a suspected/proven diagnosis of ICL.

The aim of the study will be to

1. identify patients in whom the diagnosis of ICL is confirmed using an algorithm developed by a group of multidisciplinary experts.
2. describe and compare clinical, immunological and follow up characteristics of patients in whom the diagnosis of ICL was confirmed vs patients in whom the diagnosis of ICL is not confirmed.

The investigators will also investigate :

Lymphocyte subpopulations including analysis of differentiation and activation of T and B lymphocytes, immortalisation of cell lineages with virus Epstein Barr virus, high rate genome wide genetic screening, investigation of mutations associated with identified primary immune deficiencies (adenosine deaminase et class II MHC), constitution of a biobank of frozen plasma and serum samples ; investigation of the thymic volume by performing a CT scan.

Depending on clinical presentation and based on previous data obtained by our group, the investigators will investigate the immune responses against Human papilloma virus (HPV), Cryptococcus neoformans,implication of chemokines involved in lymphocyte migration (CXCR4 and CCR7 receptors) and signalisation in response to cytokines controlling LT CD4+ homeostasis (IL-7 et IL-2).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic CD4 lymphocytopenia defined as absolute CD4+ T-lymphocyte count < 300/mm3 or < 20% of total T cells on more than one cell count; no evidence of infection with HIV-1/2 or human T-cell lymphotropic 1/2 (HTLV-1/2); and lack of a defined immune-deficiency disease or therapy for lymphocytopenia.
* Male and female patients can be included
* Children and adults can be included
* Hospitalized or outpatient

Exclusion Criteria:

* CD4+ lymphocytopenia due to another condition (HIV infection, sarcoidosis, malignant lymphoma).
* Ongoing treatment possibly responsible for CD4 lymphocytopenia.
* CD4+ lymphocytopenia related to primary immune deficiency
* Absence of consent, of inability to obtain informed consent from the patients or the right holders.
* Absence of affiliation to a social security regimen of the patient or the right holder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 patients will be included : 100 for which the diagnosis of ICL will be defined on a basis in international classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Idiopathic CD4+ T lymphocytopenia Diagnosis | 1 year
  Identify patients in whom the diagnosis of ICL is confirmed using an algorithm developed and applied by a multidisciplinary group of experts
Clinical, immunological and follow up characteristics of all patients | 1 year
  Describe and compare clinical, immunological and follow up characteristics of patients in whom the diagnosis of ICL was confirmed as compared to those in whom the diagnosis of ICL was not confirmed.

SECONDARY OUTCOMES:
Response to IL-2 or IL-7 treatment | 1 year
  Describe the response to IL-2 or IL-7 treatment
Incident cases of ICL in first degree relatives | 1 year
  Evaluate incident cases of ICL in first degree relatives of patients with ICL.
Thymic volume and correlation with CD4+ level | 1 year
  Quantify thymic volume in patients with ICL and correlate it with CD4+ level.
Analysis of differentiation and activation of T and B lymphocytes | 1 year
  Immortalisation of cell lineages with virus Epstein Barr virus, high rate genome wide genetic screening, investigation of mutations associated with identified primary immune deficiencies (adenosine deaminase et class II MHC), constitution of a biobank of frozen plasma and serum samples ; investigation of the thymic volume by performing a CT scan.
  Depending on clinical presentation and based on previous data obtained by our group, we will investigate the immune responses against Human papilloma virus (HPV), Cryptococcus neoformans,implication of chemokines involved in lymphocyte migration (CXCR4 and CCR7 receptors) and signalisation in response to cytokines controlling LT CD4+ homeostasis (IL-7 et IL-2).

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France